CLINICAL TRIAL: NCT00254436
Title: A Double-Blind, Randomized, Placebo-Controlled Study of the Efficacy and Safety of Epoetin Alfa Administered Weekly in Patients With Gastric or Rectal Cancers Undergoing Preoperative Chemoradiation Followed by Surgery
Brief Title: A Double-Blind, Randomized, Placebo-Controlled Study of the Efficacy and Safety of Weekly Procrit Given to Gastric or Rectal Patients
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Ortho Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: ID00-264
Record Dates: First submitted 2005-11-14; First posted 2005-11-16 (Estimated); Last update posted 2018-10-25 (Actual); Status verified 2018-10

CONDITIONS: Gastrointestinal Cancer; Rectal Cancer
Keywords: Epoetin Alfa; Epogen; Erythropoietin
MeSH Terms: conditions — Gastrointestinal Neoplasms; Rectal Neoplasms | interventions — Epoetin Alfa; Erythropoietin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Epoetin Alfa (Experimental)
  Interventions: Drug: Procrit (epoetin alfa)

INTERVENTIONS:
Drug: Procrit (epoetin alfa) — Weekly dose
  Other Names: Epogen; Erythropoietin

SUMMARY:
To demonstrate the effectiveness of epoetin alfa on reduction in red blood cell transfusions in gastric and rectal cancer patients undergoing preoperative chemoradiation therapy followed by surgery.

DETAILED DESCRIPTION:
Anemia and fatigue are common problems in gastric and rectal cancer subjects at the completion of chemoradiation therapy and surgery. Results of several studies in cancer subjects suggest that treatment with epoetin alfa may be effective in maintaining hemoglobin levels, thereby reducing fatigue, decreasing transfusion requirement, and potentially improving quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18 years of age or older
* Must have a confirmed diagnosis of gastric or rectal cancer for whom the treatment plan is preoperative chemoradiation followed by surgery
* Must have a baseline hemoglobin >/= 10 g/dl and < 15 g/dl
* Must have adequate hematologic function
* Must have life expectancy of more than 6 months
* Karnofsky performance status of at least 50%
* Must have adequate renal function
* Patients with reproductive potential must use an adequate contraceptive method during treatment and three months after completing treatment
* Patients must be able to read, understand, and complete the three Quality of Life questionnaires in English.

Exclusion Criteria:

* Prior chemotherapy for patients with rectal cancer
* Gastric cancer patients who have received more than 2 cycles of chemotherapy
* Anemia due to factors other than cancer/chemotherapy
* Patients with prior treatment with epoetin alfa or any investigational forms of erythropoietin within the previous 6 months
* Known hypersensitivity to mammalian-cell derived products or to human albumin
* Pregnant or lactating women
* Untreated Central Nervous System metastases
* Any significant, uncontrolled disease/dysfunction of any of the major organs
* Uncontrolled hypertension or history of uncontrolled cardiac arrhythmias, pulmonary embolism, thrombosis
* New onset or poorly controlled seizures
* History of active second malignancy
* Major infection requiring hospitalization and antibiotics or surgery within 14 days of study entry
* Blood transfusion within 1 month of study entry
* Androgen therapy within 2 months of study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2001-10-31 (Actual); Primary Completion 2004-06-29 (Actual); Study Completion 2004-06-29 (Actual)

PRIMARY OUTCOMES:
Number of Patients with Reduction in Red Blood Cell Transfusions | 2 years
Patient Iron Levels | Every 4 weeks
  Iron stores drawn at baseline and every four weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Saroj Vadhan-Raj, M.D., Principal Investigator — UT MDAnderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org